CLINICAL TRIAL: NCT00265200
Title: Bone Metabolic Markers, TRAP, and Zometa's Effect on Bone Metastasis Due to Lung Cancer
Brief Title: Using TRAP to Evaluate the Effect of Zometa on Bone Metastasis Due to Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding discontinued by sponsor
Sponsor: University of Louisville (Other)
Collaborators: James Graham Brown Cancer Center (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Goetz Kloecker, Assoc Professor, James Graham Brown Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 565.04; BCC-LUN-04-002 (Other: James Graham Brown Cancer Center Clinical Trials Office)
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Carcinoma, Non-Small Cell Lung; Carcinoma, Small Cell Lung; Metastases
Keywords: Zometa; bone metastasis; lung cancer; non-small cell lung cancer; small cell lung cancer; bone metabolic markers; tartrate resistant acid phosphatase
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Neoplasm Metastasis; Lung Neoplasms | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- zoledronic acid (Experimental): 3.0-4.0 mg by IV (in the vein), once a month for 6 months
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid — 3.0-4.0 mg by IV (in the vein), once a month for 6 months
  Other Names: Zometa

SUMMARY:
The purpose of this study is to evaluate a new blood test as a way to follow the effect of Zometa in treating bone metastases due to lung cancer.

DETAILED DESCRIPTION:
The purpose of this research study is to evaluate a new blood test as a way to follow the effect of Zometa in treating bone metastases. The blood test will look for a protein, called TRAP, which is released into the blood stream by the breakdown of bone. This study will compare the TRAP blood test with other blood tests for bone destruction.

ELIGIBILITY:
Inclusion Criteria:

* invasive lung cancer (small cell or non-small cell lung cancer)
* osteolytic bone metastasis determined by clinical exam, bone scan/XR
* age > 18 years

Exclusion Criteria:

* concurrent malignancy with a second primary
* renal failure (serum creatinine > 3mg/dl)
* pregnancy
* active rheumatoid arthritis
* intolerance to zoledronic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2005-02; Primary Completion 2009-08 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Goetz H Kloecker, MD, MSPH, Principal Investigator — James Graham Brown Cancer Center/ University of Louisville
Locations (1):
- James Graham Brown Cancer Center, Louisville, Kentucky, United States

REFERENCES:
- See also: James Graham Brown Cancer Center — http://www.browncancercenter.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zoledronic Acid
Started | 28
Completed | 24
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Average Percent Change From Baseline in TRAP Levels at 2 Weeks
Description: Change was calculated as 100% (value at baseline minus value at 2 weeks)/value at baseline
Time Frame: TRAP levels at Baseline and 2 weeks after first Zometa infusion
Population: 13 of 28 total study participants could not be evaluated: 7 due to sample deterioration; 5 participant non-compliance; 1 withdrew.
Measure: Mean (Full Range); unit: Percent change
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 15
Percent change
  NTx | 37.3 [37 to 38]
  TRAP-5b | 44.9 [44 to 45]
  bALP | 12.9 [12 to 13]

ADVERSE EVENTS:
Arm/Group | Zoledronic Acid
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes